CLINICAL TRIAL: NCT06705205
Title: Short, Animated Storytelling Video to Reduce Addiction Stigma: Protocol for a Multi-country, Online, Randomized, Controlled Trial With 13,500 Participants
Brief Title: Short, Animated Storytelling (SAS) for Addiction Stigma Reduction
Acronym: SAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Alexander von Humboldt Association (Other); Stanford Center for Digital Health (Unknown)
Responsible Party: Principal Investigator, Maya Adam, Clinical Associate Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 76457
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Social Stigma Towards People With Addiction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAS video full intervention group (Experimental): Participants view the full SAS video intervention with sound on Day 1.
  Interventions: Other: SAS video
- SAS video partial intervention (without sound) (Experimental): Participants view the partial SAS video intervention without sound on Day 1.
  Interventions: Other: SAS video
- Active Control Group (No Intervention): Participants read written information about addiction prevalence

INTERVENTIONS:
Other: SAS video — The intervention is a short, animated storytelling video, with soundtrack, aimed at reducing addiction stigma.
  Other Names: short animated storytelling video
  Arms: SAS video full intervention group; SAS video partial intervention (without sound)

SUMMARY:
Stigma towards people with addiction is a well-documented problem that negatively impacts help-seeking, treatment and recovery. Social contact with people recovering from addiction can promote empathy and reduce stigma, but social contact is difficult to scale. Short, animated storytelling (SAS) is a novel health communication approach that scales easily because it can leapfrog barriers associated with language, culture, literacy and education levels. This study will investigate if a SAS video intervention can be used to reduce stigma, boost optimism and hope, and increasing empathy towards people with addiction. The study will also explore mechanisms of action of SAS interventions, by measuring the contribution of sound design to the effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults with basic English proficiency between the ages of 18-49

Exclusion Criteria:

* None

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13397 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Addiction Stigma Scale Score as measured by the Attribution Questionnaire (AQ) | Immediately post-intervention on Day 1 and after two weeks
  Participants complete an 18-item shortened version of the validated AQ. The AQ-18 will be scored along a 9-point Likert scale indicating the extent to which participants agree with the item ranging from "not at all" to "very much" with a maximum score of 27 for each 3-item construct. Higher scores indicate greater stigma.

SECONDARY OUTCOMES:
Change in Optimism Scale Score | Immediately post-intervention on Day 1 and after two weeks
  Participants complete the Brief García's Interactive Optimism Scale (BIOS-G). The BIOS-G is an instrument designed to assess an individual's level of general optimism towards their life and other people. The scale includes 4 statements for which respondents indicate their level of agreement from 1 ("Of course not") to 4 ("Yes, of course"). Higher scores indicate a greater level of optimism.
Change in Attitude Thermometer Score | Immediately post-intervention on Day 1 and after two weeks
  Participants will indicate their warmth towards subject using a self-report stigma thermometer. Using a scale scores from zero to 100, with higher scores indicating more empathy or more favorable attitudes.
Change in Levels of Hope using a visual analogue scale (VAS) | Immediately post-intervention on Day 1 and after two weeks
  Participants self-report levels of hope using a VAS, a longstanding, validated tool for assessing related constructs of stress and subjective well-being. The scale goes from zero to 100 and higher scores indicate higher levels of hope.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Adam, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available via the Stanford Medicine Research Repository.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Adam M, Klapow M, Greuel M, Seeff M, Rohr JK, Gordon A, Amsalem D, Barnighausen T. Short, Animated Storytelling Video to Reduce Addiction Stigma in 13,500 Participants Across Multiple Countries Through an Online Approach: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 5;14:e73382. doi: 10.2196/73382. PMID 40324168